CLINICAL TRIAL: NCT03531866
Title: Web-based Resource for Youth About Clinical Research
Brief Title: Evaluation Study of Web-based Resource for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Parker, Research Scientist II, Innovation Research & Training
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHSN268201700010C
Record Dates: First submitted 2018-05-07; First posted 2018-05-22 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Chronic Disease; Healthy
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Version A (Experimental): Youth will be asked to complete a version of DigiKnowIt News that includes investigations, comics, and spotlight videos that focus on four topic areas related to participating in clincial trials. Version A will include an additional topic area.
  Interventions: Behavioral: DigiKnowIt News
- Intervention Version B (Experimental): Youth will be asked to complete a version of DigiKnowIt News that includes investigations, comics, and spotlight videos that focus on four topic areas related to participating in clincial trials. Version B will include an additional topic area (different than in Version A).
  Interventions: Behavioral: DigiKnowIt News
- Wait-List Control (No Intervention): Youth will not have access to DigiKnowIt News until after the post-test timepoint.

INTERVENTIONS:
Behavioral: DigiKnowIt News — DigiKnowIt News is an online, interactive, multimedia web-based resource designed to educate youth about participating in clinical trials. Youth will learn general information about clinical trials, their rights in a clinical trial, the good and not so good of participating in clinical trials, communication with others during a clinical trial, and specific types of procedures used in clinical trials (i.e., needles, scans). DigiKnowIt News is web-based and youth can complete it at home, on their own time.
  Arms: Intervention Version A; Intervention Version B

SUMMARY:
This study will evaluate DigiKnowIt News, a web-based resource to educate youth about pediatric clinical research. Youth will be randomly assigned to one of three groups (1. Intervention Version A; 2) Intervention Version B; 3) Wait-list control).

DETAILED DESCRIPTION:
Compared to the high numbers of clinical trials with adults, there are far fewer clinical trials with children and adolescents; highlighting the need for more clinical trials with pediatric populations. Lacking in the area of pediatric clinical research are resources to educate children and adolescents about clinical research in fun, interactive, and developmentally appropriate ways. Thus, a web-based resource, DigiKnowIt News, was developed for youth aged 8 to 14 years to educate youth about participating in pediatric clinical trials. The web-based resource includes video spotlights, investigations, and electronic comic books. The purpose of this study is to conduct a randomized controlled trial to determine the effectiveness of the web-based resource and examine its impact on youths' knowledge about pediatric clinical trials, self-efficacy about making decisions about participation in clinical research, and positive attitudes towards participation.

ELIGIBILITY:
Inclusion Criteria:

* Within the ages of 8 and 14 years of age

Exclusion Criteria:

* Does not speak English fluently, does not have access to a computer or tablet with internet connection, and or has participated in a clinical trial after kindergarten.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge about Clinical Research | 2 weeks
  Questions will assess youth's factual knowledge about clinical research using a multiple choice format.
Change in Attitudes toward Clinical Research | 2 weeks
  Questions will assess youth's attitudes toward pediatric clinical research on a 3-point Likert rating scale.
Change in Self-Efficacy for Making Decisions | 2 weeks
  Questions will assess youth's self-efficacy for making decisions using a 5-point Likert scale.

SECONDARY OUTCOMES:
Changes in Initiative-Taking | 2 weeks
  Questions will assess youth's initiative-taking using a 5-point Likert scale.
Changes in Hope | 2 weeks
  Questions will assess youth's perceptions of hope using a 6-point Likert scale.
Changes in Parent-Child Communication | 2 weeks
  Questions will assess youth's perceptions about the quality of communication in their parent-child relationship using a 5-point Likert scale.
Consumer Satisfaction | 1 day
  Questions will ask youth to reflect on their experiences with the web-based resource using 5-point Likert scales.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Parker, PhD, Principal Investigator — Innovation Research & Training; Tracy Scull, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No